CLINICAL TRIAL: NCT07331909
Title: Assessing the Use of Wearable Activity Trackers in a Pregnancy Cohort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Danielle Prentice, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00028457
Record Dates: First submitted 2025-11-25; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related
Keywords: Wearable Activity Tracker

STUDY DESIGN:
Intervention Model Description: All participants will wear the Garmin Vivosmart 5 wearable activity tracker. Participants will be randomized 1:1 to whether they have access to their activity data from the tracker or if they are blinded to their activity tracker.
Masking Description: Participants and research team members will know which arm participants in. Participants in the blinded arm will not have access to their data from the wearable activity tracker.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable Activity Tracker with Data Access (Experimental): Participants will wear a Garmin Vivosmart 5 wearable activity tracker and have access to the data it collects.
  Interventions: Device: Wearable Activity Tracker
- Blinded Wearable Activity Tracker (No Intervention): Participants will wear a Garmin Vivosmart 5 wearable activity tracker and be blinded to the data it collects.

INTERVENTIONS:
Device: Wearable Activity Tracker — A watch-style wearable activity tracker which tracks steps, heart rate, activity level, and sleep quality.
  Other Names: Garmin Vivosmart 5
  Arms: Wearable Activity Tracker with Data Access

SUMMARY:
This is a randomized controlled pilot study to evaluate the utility of the Garmin Vivosmart 5 wearable activity tracker in pregnancy. It will determine the feasibility of assessing physical activity in pregnant patients using wearable activity trackers and collect pilot data on the behavioral impact of wearable activity trackers on physical activity in pregnancy.

DETAILED DESCRIPTION:
Pregnant participants will be given a Garmin Vivosmart 5 wearable activity tracker. They will be randomized 1:1 as to whether they are able to see their personal activity information or being blinded to it. Participants will complete a questionnaire on their physical activity levels before initiating use of the activity tracker and following delivery. Participants' physical activity data, satisfaction with the device, and gestational and delivery outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Establishing pregnancy care at Oregon Health & Science University
* Gestational age less than or equal to 24 weeks and 6 days
* Ability to read, write and speak English
* Ability to upload data either at home via a stable internet connection or in clinic

Exclusion Criteria:

* Non-English speaking
* Inability to wear wearable fitness technology due to allergy or sensory issues
* Inability to upload data from wearable fitness technology due to lack of stable internet connection or ability to come to clinic for upload via the research team in the timeframe required
* Inability to answer electronic questionnaires
* Specific contraindication to increased physical activity in pregnancy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Device use | Measured from study enrollment through 6 weeks postpartum, an average of 26 weeks
  The number of days that participants wear the study device during the study period
Participant satisfaction | Measured at 6 weeks postpartum.
  Participant survey question asking "On a scale of 1 to 100, how satisfied were you with the activity tracker?" With a higher value representing a greater degree of satisfaction.

SECONDARY OUTCOMES:
Physical activity | From enrollment through delivery
  The mean number of minutes of physical activity per week recorded by the wearable activity tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Prentice, DO, Principal Investigator — Oregon Health and Science University